CLINICAL TRIAL: NCT03715439
Title: Evaluation of Dental Implants Placed in Preserved Post-extraction Ridges With Leucocyte- and Platelet-rich Fibrin: 1, 3 and 5-year Post-loading Outcome of a Randomized Controlled Trial
Brief Title: Evaluation of Dental Implants Placed in Preserved and Non-preserved Post-extraction Ridges
Status: Withdrawn | Type: Observational
Why Stopped: Duo to pandemic period (COVID) the surgical elective procedures were stopped
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, João Vitor dos Santos Canellas, DDS MS, DDS MS, Rio de Janeiro State University
Other Study IDs: 72596717.3.0000.5259/2
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Dental Implant Failed; Platelet-rich Fibrin; Alveolar Rege Preservation; Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Leucocyte- and Platelet-rich Fibrin: Dental implant placed into post-extraction sites preserved with leucocyte- and platelet-rich fibrin
  Interventions: Device: Dental implant
- Control: Dental implant placed into non-preserved post-extraction sites
  Interventions: Device: Dental implant

INTERVENTIONS:
Device: Dental implant — A single dental implant was inserted 3 months after tooth extraction

SUMMARY:
A prospective study to evaluate and compare implants placed in preserved versus non-preserved extraction sockets using L-PRF (Leucocyte- and platelet-rich fibrin) after 1, 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Health patients, American Society of Anesthesiologists (ASA) I or II
* Patients who need to submit tooth extraction (pre-molar, canine and incisor teeth which present ideal conditions to receive dental implants after 3 months.

Exclusion Criteria:

* Systemic diseases related with healing disorders
* Poor oral hygiene
* Pregnant or lactating patient
* Use of flap elevation for dental extraction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study presents the 1,3 and 5-year evaluation of a previously accomplished randomized, clinical study initiated in 2018. The study sample was recruited among patients referred to the School of Dentistry, University of Rio de Janeiro, Brazil for treatment with single-tooth implants.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
survival rates of the implants | 1 year
  The term surviving refers to those implants that are still in the jaw of the patient but either have not met success criteria or have not been tested for success.
survival rates of the implants | 3 years
  The term surviving refers to those implants that are still in the jaw of the patient but either have not met success criteria or have not been tested for success.
survival rates of the implants | 5 years
  The term surviving refers to those implants that are still in the jaw of the patient but either have not met success criteria or have not been tested for success.
success rates of the implants | 1 year
  Success is graded in three qualities, depending on the extent and results of performed examinations.
  Grade 1.
  1. Absence of mobility is checked by individual stability testing of the unattached implant.
  2. Radiographic evaluation of each implant reveals not more than 1.0 mm of marginal bone loss during the first year of loading, followed by not more than 0.2 mm resorption per year.
  3. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc.
  Grade 2.
  1. Radiographic evaluation
  2. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc, are absent.
  Grade 3.
  1. Radiographic evaluation. Peri-implant pathosis, such as a peri-implant radiolucency is absent.
  2. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc, are absent.
success rates of the implants | 3 years
  Success is graded in three qualities, depending on the extent and results of performed examinations.
  Grade 1.
  1. Absence of mobility is checked by individual stability testing of the unattached implant.
  2. Radiographic evaluation of each implant reveals not more than 1.0 mm of marginal bone loss during the first year of loading, followed by not more than 0.2 mm resorption per year.
  3. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc.
  Grade 2.
  1. Radiographic evaluation
  2. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc, are absent.
  Grade 3.
  1. Radiographic evaluation. Peri-implant pathosis, such as a peri-implant radiolucency is absent.
  2. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc, are absent.
success rates of the implants | 5 years
  Success is graded in three qualities, depending on the extent and results of performed examinations.
  Grade 1.
  1. Absence of mobility is checked by individual stability testing of the unattached implant.
  2. Radiographic evaluation of each implant reveals not more than 1.0 mm of marginal bone loss during the first year of loading, followed by not more than 0.2 mm resorption per year.
  3. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc.
  Grade 2.
  1. Radiographic evaluation
  2. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc, are absent.
  Grade 3.
  1. Radiographic evaluation. Peri-implant pathosis, such as a peri-implant radiolucency is absent.
  2. Severe soft tissue infections, persistent pain, paresthesia, discomfort, etc, are absent.

SECONDARY OUTCOMES:
Marginal Bone Loss | 1 year
  Periapical digital radiographs will be used to make the measurements and evaluations.
Marginal Bone Loss | 3 years
  Periapical digital radiographs will be used to make the measurements and evaluations.
Marginal Bone Loss | 5 years
  Periapical digital radiographs will be used to make the measurements and evaluations.
Pink Esthetic Score | 1 year
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
Pink Esthetic Score | 3 years
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
Pink Esthetic Score | 5 years
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
Patient satisfaction - Questions will be scored on 100mm visual analog scales. The patients marked their response on a horizontal line for which the most negative expression corresponded to 0 and the most positive to 100. | 1 year
  Questions: Are you satisfied with the aesthetic outcome of the gums surrounding this implant? Are you satisfied with the function of your implant-supported tooth? Would you undergo the same procedure again?
Patient satisfaction - Questions will be scored on 100mm visual analog scales. The patients marked their response on a horizontal line for which the most negative expression corresponded to 0 and the most positive to 100. | 3 years
  Questions: Are you satisfied with the aesthetic outcome of the gums surrounding this implant? Are you satisfied with the function of your implant-supported tooth? Would you undergo the same procedure again?
Patient satisfaction - Questions will be scored on 100mm visual analog scales. The patients marked their response on a horizontal line for which the most negative expression corresponded to 0 and the most positive to 100. | 5 years
  Questions: Are you satisfied with the aesthetic outcome of the gums surrounding this implant? Are you satisfied with the function of your implant-supported tooth? Would you undergo the same procedure again?
Patient satisfaction with single-tooth implant treatment measured with the Oral health impact profile-14 questionnaire | 1 year
  The questionnaire was divided into seven domains, containing two questions each, resulting in a total of 14 questions. The domains were functional limitation physical disability, physical pain, psychological disability, psychological discomfort, social disability and handicap. The overall OHIP-14 score is the mean of the 14 questions. The questions pertained to seven domains and were averaged on a scale of 0-4, with 0 defined as "never" a problem and 4 defined as "very often" a problem.
Patient satisfaction with single-tooth implant treatment measured with the Oral health impact profile-14 questionnaire | 3 years
  The questionnaire was divided into seven domains, containing two questions each, resulting in a total of 14 questions. The domains were functional limitation physical disability, physical pain, psychological disability, psychological discomfort, social disability and handicap. The overall OHIP-14 score is the mean of the 14 questions. The questions pertained to seven domains and were averaged on a scale of 0-4, with 0 defined as "never" a problem and 4 defined as "very often" a problem.
Patient satisfaction with single-tooth implant treatment measured with the Oral health impact profile-14 questionnaire | 5 years
  The questionnaire was divided into seven domains, containing two questions each, resulting in a total of 14 questions. The domains were functional limitation physical disability, physical pain, psychological disability, psychological discomfort, social disability and handicap. The overall OHIP-14 score is the mean of the 14 questions. The questions pertained to seven domains and were averaged on a scale of 0-4, with 0 defined as "never" a problem and 4 defined as "very often" a problem.

CONTACTS AND LOCATIONS:
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided